CLINICAL TRIAL: NCT00378911
Title: A Phase II Evaluation of Sunitinib Malate (Sutent®, SU11248, NCI-Supplied Agent , NSC # 736511) in the Treatment of Recurrent or Persistent Leiomyosarcoma of the Uterus
Brief Title: Sunitinib in Treating Patients With Recurrent or Persistent Leiomyosarcoma of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02702; NCI-2012-02702 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000495190; GOG-0231C (Other: Gynecologic Oncology Group); GOG-0231C (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Uterine Sarcoma; Uterine Leiomyosarcoma
MeSH Terms: interventions — Sunitinib

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with recurrent or persistent leiomyosarcoma of the uterus. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the activity of sunitinib malate, in terms of rate of progression-free survival for ≥ 6 months and objective tumor response, in patients with recurrent or persistent leiomyosarcoma of the uterus who have received 1 or 2 prior cytotoxic therapies.

II. Determine the frequency and severity of adverse events.

SECONDARY OBJECTIVES:

I. Determine the duration of progression-free survival and overall survival.

OUTLINE: This is a multicenter study. Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed leiomyosarcoma of the uterus

  * Recurrent or persistent disease
  * Refractory to curative therapy or established treatments
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan

  * Ascites and pleural effusions are not considered measurable disease
* Must have ≥ 1 target lesion to assess response

  * Tumors in a previously irradiated field are considered non-target lesions unless there is documented progression or biopsy-confirmed persistence ≥ 90 days after completion of radiotherapy
* Received at least 1 but no more than 2 prior cytotoxic regimens

  * Initial treatment may have included high-dose chemotherapy, consolidation, or extended therapy administered after surgery or nonsurgical assessment
  * Cytotoxic regimens may have included any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
* Not a candidate for a higher priority GOG protocol
* No known brain metastases
* GOG performance status 0-2 (for patients who have received 1 prior regimen) OR GOG 0-1 (for patients who have received 2 prior regimens)
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* QTc < 500 msec
* LVEF normal by echocardiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 1 month after completion of study treatment
* Patients with a pre-existing thyroid abnormality unable to maintain normal thyroid function with medication are not eligible
* No significant EKG abnormalities (i.e., no history of serious ventricular arrhythmia OR EKG with ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No sensory or motor neuropathy > grade 1
* No NYHA class III-IV congestive heart failure

  * NYHA class II cardiac dysfunction allowed
  * History of NYHA class II heart failure that is asymptomatic on treatment allowed
* No active infection requiring antibiotics
* No other invasive malignancies within the past 5 years except for nonmelanoma skin cancer
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib malate
* No poorly controlled hypertension (i.e., systolic blood pressure [BP] ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg)
* No gastrointestinal tract disease resulting in an inability to take oral medication
* No requirement for IV alimentation
* No active peptic ulcer disease
* No other condition that would impair ability to swallow and retain study drug
* No serious or nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No cerebrovascular accident or transient ischemic attack within the past year
* No myocardial infarction, cardiac arrhythmia, stable or unstable angina, or symptomatic congestive heart failure within the past year
* No pulmonary embolism within the past year
* No uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infections
  * Psychiatric illness or social situations that would preclude study compliance
* Recovered from prior surgery, chemotherapy, or radiotherapy
* Prior anthracycline exposure and central thoracic radiation that included the heart allowed provided patient has New York Heart Association (NYHA) class II cardiac function
* At least 1 week since prior hormonal therapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin C) or radiotherapy
* At least 4 weeks since prior major surgery
* At least 3 years since prior radiotherapy for localized cancer of the breast, head and neck, or skin and no recurrent or metastatic disease
* At least 3 years since prior adjuvant chemotherapy for localized cancer of the breast and no recurrent or metastatic disease
* No prior radiotherapy to any portion of the abdominal cavity or pelvis unless for treatment of leiomyosarcoma
* No prior chemotherapy to any portion of the abdominal cavity or pelvis unless for treatment of leiomyosarcoma
* No prior noncytotoxic chemotherapy for recurrent or persistent disease
* No prior surgical procedures affecting absorption
* No coronary or peripheral artery bypass graft or stenting within the past year
* No other prior antiangiogenic agents (e.g., bevacizumab, sorafenib, pazopanib, AZD2171, vatalanib, or vascular endothelial growth factor [VEGF] Trap)
* No other prior cancer treatment that would preclude study treatment
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * Azole fungals (e.g., ketoconazole or itraconazole)
  * Clarithromycin
  * Erythromycin
  * Diltiazem
  * Verapamil
  * HIV protease inhibitors (e.g., indinavir, saquinavir, ritonavir, atazanavir, or nelfinavir)
  * Delavirdine
* At least 12 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * Hypericum perforatum (St. John's wort)
  * Efavirenz
  * Tipranavir
* No concurrent proarrhythmic potential agent, including any of the following:

  * Terfenadine
  * Quinidine
  * Procainamide
  * Disopyramide
  * Sotalol
  * Probucol
  * Bepridil
  * Haloperidol
  * Risperidone
  * Indapamide
  * Flecainide
* No concurrent therapeutic coumarin-derivative anticoagulants, such as warfarin

  * Doses ≤ 2 mg daily allowed for prophylaxis of thrombosis
  * Low molecular weight heparin allowed provided PT INR ≤ 1.5
* No concurrent amifostine or other protective agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From study entry until disease progression, death or date of last contact., assessed up to 6 months
Objective tumor response according to GOG RECIST criteria | Up to 5 years
Frequency and severity of adverse events as assessed by CTCAE v 3.0 | Up to 5 years
  The frequency and severity of all toxicities will be tabulated.

SECONDARY OUTCOMES:
Duration of progression-free survival | Up to 5 years
  Characterized graphically and using descriptive statistics such as median survival.
Duration of overall survival | From entry into the study to death or the date of last contact, assessed up to 5 years
  Characterized graphically and using descriptive statistics such as median survival.

CONTACTS AND LOCATIONS:
Overall Officials: Martee Hensley, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States